CLINICAL TRIAL: NCT02846272
Title: Diffusion Tensor and Functional Connectivity Imaging in Pediatric Epilepsy: Imaging/Histology Correlation
Acronym: DTI/SEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Manish Narendra Shah, M.D. , Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-15-0022
Record Dates: First submitted 2016-07-08; First posted 2016-07-27 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Intractable Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observational cohort (Experimental): Observing MRI changes in subjects.
  Interventions: Procedure: Observation

INTERVENTIONS:
Procedure: Observation — Observation of MRI changes in subjects

SUMMARY:
To determine the utility of diffusion tensor magnetic resonance imaging in the preoperative workup of children with intractable epilepsy referred for surgery.

DETAILED DESCRIPTION:
To determine if diffusion tensor and functional connectivity magnetic resonance imaging helpful to better understand and diagnose intractable epilepsy in children. All enrolled children will undergo standard preoperative and postoperative MRI imaging, plus a 15 minute set of functional connectivity and diffusion tensor sequence with no additional sedation. This imaging data will be stripped of identifiers and be processed to provide both quantitative analysis, resting state functional connectivity changes and three dimensional modeling of white matter tracts adjacent to epileptogenic foci. This study is being done to determine if diffusion tensor and functional connectivity magnetic resonance imaging are helpful to better understand and diagnose intractable epilepsy in children.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosis with Intractable Epilepsy

Exclusion Criteria:

* No Intractable Epilepsy

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with seizure outcome as determined by Engel | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Manish N Shah, M.D., Principal Investigator — UTHealth Medical School
Locations (1):
- UTHealth & Children's Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No